CLINICAL TRIAL: NCT02154841
Title: Changes in Taste Perception and Preference in the Peri-operative Patient
Acronym: TASTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11/P/009; 10/H0203/74 (Other: National Research Ethics Service)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Post Operative Nutrition
Keywords: Postoperative; nutrition; taste; perception; preference; choice
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Questionnaire, taste test, visual food test (Experimental): The participants will complete a questionnaire that asks them about their taste preferences. They will also will be shown photos of various food stuffs and asked to choose their preferred meal. They will also be asked to put five sponge sticks (a single use item commonly used for mouth care) dipped in one of a five different liquids into their mouths and give their comments what each taste was and on how much they enjoyed it. These five liquids represent the four well-described tastes (sweet, sour, salty, bitter) and a more recently proposed taste, savoury. The intention of this part of the trial is to assess the patient's ability to detect alteration in pure taste and to identify if any of these tastes are preferred.
  Interventions: Behavioral: Questionnaire, taste test, visual food test

INTERVENTIONS:
Behavioral: Questionnaire, taste test, visual food test

SUMMARY:
It is well known that patients who have undergone major surgical procedures are vulnerable to the consequences of inadequate calorie or nutritional intake. Clinical studies have demonstrated that early post-operative feeding increases strength and healing of an intestinal anastomosis, reduces surgical site infection and length of hospital stay. The 'Enhanced recovery programme', ERP, includes early post-operative nutrition as one of its key goals, however there is no guidance on the type of food that should be offered to patients in this programme. Anecdotally, many patients and healthcare professionals believe that there are differences in how food tastes to early post-operative patients. If there are changes in taste following surgery this will affect the food choices that patients make in the early post-operative period. No studies have addressed this question to date. In this study we hope to describe this affect and consider the significance of any changes on the background of current hospital food options.

We hypothesise that food preference and tastes and desires are altered in the early post operative period and this affects what patients eat at this critical time.

DETAILED DESCRIPTION:
Nutrition is a vital component of good health and recovery from illness. It is particularly clear that patients with chronic diseases and those who have undergone major surgical procedures are vulnerable to the consequences of inadequate calorie or nutritional intake. Over the last decade, surgical practices have evolved to encourage patients to resume early enteral feeding in order to avoid post-operative under-nutrition. Inadequate nutrition has previously been shown to be associated with prolongation of the acute phase response and increased incidence of septic morbidity. More recently clinical studies have demonstrated that early post-operative feeding increases strength and healing of an intestinal anastomosis. Further to this there is also evidence of benefit to patients by reduction of surgical site infections and other complications. Along with the cost saving of a lower complication rate there are financial benefits from reduced mean length of hospital stay.

Over the last 5 years the importance of non-surgical factors in patient recovery or the development of complications has been highlighted. This has resulted in the development and near universal adoption of the 'Enhanced recovery programme (ERP)'. The ERP is a multidisciplinary initiative aiming to improve the patients' journey by:

* Optimizing pre-operative health status
* Reducing postoperative complications and the surgical and physiological stress responses by changing traditional surgical methods
* Early mobility
* Early feeding Post-operative nutrition is a key component to the ERP approach, however, many units that run ERP have reported that encouraging early post operative patients to increase their oral intake is difficult. Our own experience is that dysgeusia (distortion of the sense of taste) is common in the postoperative group.

At present there are no publications in the literature on how best to support the delivery of nutrition to this important group and there is no literature on food preferences in patients who have recently undergone surgery. To date there has not been any research on the subject of peri-operative taste changes outside of surgical fields that directly affect the sensory system of taste (Ear, nose and throat surgery). Although there have been some descriptive studies on calorie intake in the peri-operative period no studies have been performed to confirm the existence of post-operative taste changes or to describe them.

In order to optimise recovery from surgery and as part of the ERP programme, patients should be provided with food choices that encourage greater intake. It is known that optimising early post-operative nutrition will contribute to early discharge and uncomplicated recovery and have knock on benefits for inpatient costs. In order to provide this it is vital that we consider the issue of presumed dysgeusia and its affect on food choices. In order to begin this process the following study is proposed. It is hoped that the results of this study will allow re-evaluation of hospital menus to optimise post-operative nutrition.

ELIGIBILITY:
Inclusion Criteria:

Patients who undergo the following laparoscopic procedures

* anterior resection
* right/Left hemicolectomy
* sigmoid colectomy
* abdominal-perineal resection
* stoma formation

Exclusion Criteria:

The participant may not enter the study if:

* patients under 18 years old
* if they report any protracted change in taste over the 6 months prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To describe taste appreciation and detection in the pre and post-operative Assess taste changes in the peri-operative patient | 3 days post operation
  Patients that agree to participate will complete a questionnaire that asks them about their taste preferences. Recruits will be shown photos of various food stuffs and asked to choose their preferred meal. They will also be asked to put five sponge sticks (a single use item commonly used for mouth care) dipped in one of a five different liquids into their mouths and give their comments what each taste was and on how much they enjoyed it. These five liquids represent the four well-described tastes (sweet, sour, salty, bitter) and a more recently proposed taste, savoury. The intention of this part of the trial is to assess the patient's ability to detect alteration in pure taste and to identify if any of these tastes are preferred.

SECONDARY OUTCOMES:
Assess taste preferences in the peri-operative patient | 3 days post operation
  Patients that agree to participate will complete a questionnaire that asks them about their taste preferences. Recruits will be shown photos of various food stuffs and asked to choose their preferred meal. They will also be asked to put five sponge sticks (a single use item commonly used for mouth care) dipped in one of a five different liquids into their mouths and give their comments what each taste was and on how much they enjoyed it. These five liquids represent the four well-described tastes (sweet, sour, salty, bitter) and a more recently proposed taste, savoury. The intention of this part of the trial is to assess the patient's ability to detect alteration in pure taste and to identify if any of these tastes are preferred.
Patients choice of meal from a selection of photographs of food | 3 days post operation
  Patients that agree to participate will complete a questionnaire that asks them about their taste preferences. Recruits will be shown photos of various food stuffs and asked to choose their preferred meal. They will also be asked to put five sponge sticks (a single use item commonly used for mouth care) dipped in one of a five different liquids into their mouths and give their comments what each taste was and on how much they enjoyed it. These five liquids represent the four well-described tastes (sweet, sour, salty, bitter) and a more recently proposed taste, savoury. The intention of this part of the trial is to assess the patient's ability to detect alteration in pure taste and to identify if any of these tastes are preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lewis, M.B., Ch.B., M.D., Study Director — University Hospital Plymouth NHS Trust; Sophie-Anne Welchman, B.Sc.(Hons), M.B.B.S., Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom